CLINICAL TRIAL: NCT03466697
Title: Role of Dopamine Transporter in Glucose Loading of Healthy Subjects
Brief Title: Role of Dopamine Transporter in Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Kyoungjune Pak, Clinical Assistant Professor, Pusan National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1707-019-057
Record Dates: First submitted 2018-03-08; First posted 2018-03-15 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Glucose; Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Other): All subjects will be injected twice for each visit (normal saline or glucose)
  Interventions: Other: Glucose injection/Normal saline injection

INTERVENTIONS:
Other: Glucose injection/Normal saline injection — Before each PET scan, subject will be injected either glucose or normal saline.

SUMMARY:
Healthy subjects will be enrolled in this study. Each subject will be scanned twice with F18-FP-CIT PET which is commercially available. F18-FP-CIT reflects dopamine transporter availability of striatum. Before each PET scan, subject will be injected either glucose or normal saline. Therefore, PET scan will reflect the changes of dopamine transporter availability after the injection of glucose.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* known neurologic disorder
* known drug addiction
* known endocrine disorder

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Specific binding ratio of dopamine transporter availabilitiy measured from PET scans | less than 1 month
  Specific binding ratio of dopamine transporter availabilitiy measured from PET scans

CONTACTS AND LOCATIONS:
Overall Officials: Kyoungjune Pak, MD, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No